CLINICAL TRIAL: NCT03691506
Title: Comparison of Constraint-induced Movement Therapy and Its Modified Form on Upper Motor Function Outcomes and Psychosocial Impact in Hemiplegic Cerebral Palsy.
Brief Title: Comparison of CIMT and Its Modified Form on Upper Motor Function Outcomes in Hemiplegic Cerebral Palsy.
Acronym: CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Mamoona Tasleem Afzal
Record Dates: First submitted 2018-09-14; First posted 2018-10-01 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Cerebral Palsy; Constraint-Induced Movement Therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic CIMT group (Active Comparator): Total session of 6 hours a day, 5 days per week for 3 weeks to Classic CIMT groups will be given.
  Interventions: Other: Classic CIMT group
- mCIMT group (Experimental): Session of 6 hours a day, 5 session per week for first 2 weeks (CIMT), session of 2 hours a day, 5 days per week for last 1 week (BIT) to modified CIMT group will be given.
  Interventions: Other: Modified CIMT group

INTERVENTIONS:
Other: Classic CIMT group — Constraint Induced Movement Therapy (CIMT) is a new treatment technique that claims to improve the arm motor ability and the functional use of a paretic arm - hand. CIMT forces the use of the affected side by restraining the unaffected side. Child with hemiplegic cerebral palsy can learn to improve the motor ability of the more affected parts of their bodies and thus cease to rely exclusively or primarily on the less affected parts.
  Arms: Classic CIMT group
Other: Modified CIMT group — Modified CIMT protocol that was based on suggestions made by Dromerick, Edwards, and Hahn (2000) . Modifications were reductions in the duration of mitt wear and massed practice compared with the traditional protocol
  Arms: mCIMT group

SUMMARY:
The aim of this research is to compare the effect of classic constraint-induced movement therapy and its modified form on upper extremity motor function outcomes and psychosocial impact in hemiplegic cerebral palsy. Randomized controlled trials with 2-3 weeks follow-up. The sample size is 40. The subjects are divided in two groups, 20 subjects in classical CIMT group and 20 in modified CIMT group. Study duration is of 6 months. Sampling technique applied will be purposive non probability sampling technique. Only 4-12 years individual with hemiplegic cerebral palsy are included. Tools used in the study are Box and Block test, Cerebral palsy (quality of life), Kid Screen 27 and QUEST (quality of upper extremity skill test). Data will be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Cerebral palsy is known as a neurodevelopment disease that begins in the early childhood and persists throughout the life. In the past, it was a challenge to define the term CP. Many attempts were made to overcome this. In 1964, definition for cerebral palsy was given that is still used worldwide. According to that cerebral palsy (CP) is not just the disorder of posture but movement also and it happens due to lesion or damage of an immature brain. It is a disorder of human brain that is non-progressive. The main focus of the definition was on the motor impairment. Cerebral palsy can lead to activity limitation. As CP includes motor disorders so it encounters disturbances like cognition, sensation, communication, seizures and behavioral disorder.

The frequency with which CP occurs is of importance as it is the first effort towards its prevention. It also estimates the supportive services and the medical care that is required for children with cerebral palsy and also their families. Many studies were conducted to check the trends of Cerebral Palsy occurrence depending upon the low birth weight.

The definition of cerebral palsy shows that it is just a single disorder infect it is collection of disorders. Prevalence of cerebral palsy shows that out of 1000 births, there are 2.0-2.5 children are victims of cp. However in few children, the causes of CP are still not known. Moreover, the causes need to be discriminated from the risk factors. Prenatal events are also responsible for CP. Such events may include toxins, maternal infection for example rubella or brain malformations. One of the prenatal causes is birth asphyxia. A small ratio of CP can be the result of perinatal causes. 10% cases of cp are result of postnatal causes. The causes can be accidental or non-accidental. Meningitis is also one of the postnatal causes.

Out of all types of cerebral palsy, one-third is spastic hemiplegic. Birth trauma can be the cause of spastic hemiplegia. Researches show that there is more ratio of right hemiplegia than the left hemiplegia. The most common form of CP that is seen in premature children is spastic diplegia. In spastic diplegia, spasticity affects lower limbs more than the upper extremity. Birth asphyxia is seen in children born with the choreo-athetosis.

Traditional hemiplegic patients receive occupational and physical therapy to improve their functional skills. Constraint induced movement therapy (CIMT) is an approach to treating the hemiparesis that facilitate use of hemiparetic arm through constraint the unaffected arm.it has been shown to be effective treatment in hemiparesis in adult and children.

In this study, I hypothesized that there is a difference between the effectiveness of classic CIMT with modified CIMT on upper extremity motor function outcomes in children with hemiplegic cerebral palsy. The purpose of this study is to compare the effects of classic CIMT with modified CIMT on upper extremity motor functions and to see the psychosocial impact of CIMT on hemiplegic cerebral palsy.

LITERATURE REVIEW:

There is injury of undeveloped brain in Children with CP. Children with hemiplegic cerebral palsy (HCP) have trouble using their affected arm and hand on one side of their body. Evidence from randomized controlled trials, clinical controlled trials, and systematic reviews has shown constraint therapy improves hand and arm movement in children with hemiplegic cerebral palsy. According to a research review done in 2014; it is seen that CIMT proved to be beneficial in improving hand function as compared to the conventional therapy. A comparison was done between equal intensity of bimanual training and CIMT. Results showed same progress in hand function.

A comparison was done between equal intensity of hand arm bimanual training (HABIT) and CIMT. Results showed same progress in hand function. Modified constraint-induced movement therapy improved isolated functions of the hemiplegic arm better than intensive bimanual training, but regarding spontaneous hand use in everyday life both methods lead to similar improvement. This suggests mCIMT should be paired with BIT to achieve optimal results for children with HCP who present with difficulties in both unimanual and bimanual hand functions. A study combining mCIMT and BIT demonstrated more frequent and more effective use of the affected limb, and better performance inself-care and leisure tasks.

Children and parents from both groups (CIMT and BIT) reported a significant improvement in their or their child's feelings about functioning as well as participation and physical health. The parents of children receiving CIMT reported positive and sustained changes in their child's social well-being (CPQOL-Child). The CIMT group showed significant improvements in physical well-being, psychological well-being, moods and emotions.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 12 years CP with unilateral, bilateral or severely asymmetrical impairment Manual Ability Classification System(MACS) I, II or III
* Wrist extension capacity at least 20°; fingers with 10° of complete flexion
* Children able to follow Command

Exclusion Criteria:

* Children also having disabilities other than Cerebral palsy
* Contractures that significantly limit functional arm use.
* Children with MR.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline [Box And Block Test (BBT)] at 3rd week | 3rd week
  The Box and Blocks Test (BBT) is a functional test used in upper limb rehabilitation.The test is used to measure the gross manual dexterity of a patient.The test consists of a box with a partition in the middle. Blocks are placed at one side of the partition. The box is placed at a table. The test subject is seated, facing towards the box. During the tests the test subject is given 60 seconds to move as many blocks as possible from one side to the other, by using only his tested hand. The number of displaced blocks is a measure of the gross manual dexterity. A higher number of displaced blocks indicates a better gross dexterity.

SECONDARY OUTCOMES:
Change from Baseline [Quality Of Upper Extremity Skill Test (QUEST)] at 3rd week | 3 weeks.
  The Quality of Upper Extremity Skills Test is an outcome measure designed to evaluate movement patterns and hand function in children with cerebral palsy. The QUEST is both reliable and valid. The purpose of the QUEST is to evaluate quality of upper extremity function in four domains: dissociated movement, grasp, protective extension, and weight bearing. 36 items assessing dissociated movements, grasp, protective extension, and weight bearing.
Change from Baseline [Kid Screen 27] at 3rd week | 3 weeks.
  The KIDSCREEN-27 was developed as a shorter version of the KIDSCREEN-52 with a minimum of information loss and with good psychometric properties. The KIDSCREEN-27 with five dimensions resulted. All five dimensions are Rasch scales: Physical Well-Being (5 items), Psychological Well-Being (7 items), Autonomy & Parents (7 items), Peers & Social Support (4 items), and School Environment (4 items).
Change from Baseline [Cerebral Palsy Quality of Life CP(QOL)] at 3rd week | 3 weeks.
  The Cerebral Palsy Quality of Life for Children (CP QOL-Child) is the first health condition-specific questionnaire designed for measuring QOL in children with cerebral palsy (CP) aged 4-12 years. CP QOL Questionnaires measure include : Social wellbeing & acceptance, Feelings about functioning, Participation & physical health, Emotional wellbeing & self-esteem, Access to services, Pain & impact of disability, Family health.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PHD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maenner MJ, Blumberg SJ, Kogan MD, Christensen D, Yeargin-Allsopp M, Schieve LA. Prevalence of cerebral palsy and intellectual disability among children identified in two U.S. National Surveys, 2011-2013. Ann Epidemiol. 2016 Mar;26(3):222-6. doi: 10.1016/j.annepidem.2016.01.001. Epub 2016 Jan 12. PMID 26851824
- [Background] Winter S, Autry A, Boyle C, Yeargin-Allsopp M. Trends in the prevalence of cerebral palsy in a population-based study. Pediatrics. 2002 Dec;110(6):1220-5. doi: 10.1542/peds.110.6.1220. PMID 12456922
- [Background] Himmelmann K, Beckung E, Hagberg G, Uvebrant P. Gross and fine motor function and accompanying impairments in cerebral palsy. Dev Med Child Neurol. 2006 Jun;48(6):417-23. doi: 10.1017/S0012162206000922. PMID 16700930
- [Background] Reddihough D. Cerebral palsy in childhood. Aust Fam Physician. 2011 Apr;40(4):192-6. PMID 21597527
- [Background] Al-Oraibi S, Eliasson AC. Implementation of constraint-induced movement therapy for young children with unilateral cerebral palsy in Jordan: a home-based model. Disabil Rehabil. 2011;33(21-22):2006-12. doi: 10.3109/09638288.2011.555594. Epub 2011 Feb 18. PMID 21332299
- [Background] Facchin P, Rosa-Rizzotto M, Visona Dalla Pozza L, Turconi AC, Pagliano E, Signorini S, Tornetta L, Trabacca A, Fedrizzi E; GIPCI Study Group. Multisite trial comparing the efficacy of constraint-induced movement therapy with that of bimanual intensive training in children with hemiplegic cerebral palsy: postintervention results. Am J Phys Med Rehabil. 2011 Jul;90(7):539-53. doi: 10.1097/PHM.0b013e3182247076. PMID 21765273
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350
- [Background] Hoare B, Imms C, Carey L, Wasiak J. Constraint-induced movement therapy in the treatment of the upper limb in children with hemiplegic cerebral palsy: a Cochrane systematic review. Clin Rehabil. 2007 Aug;21(8):675-85. doi: 10.1177/0269215507080783. PMID 17846067
- [Background] Eliasson AC, Krumlinde-sundholm L, Shaw K, Wang C. Effects of constraint-induced movement therapy in young children with hemiplegic cerebral palsy: an adapted model. Dev Med Child Neurol. 2005 Apr;47(4):266-75. doi: 10.1017/s0012162205000502. PMID 15832550
- [Background] Tinderholt Myrhaug H, Ostensjo S, Larun L, Odgaard-Jensen J, Jahnsen R. Intensive training of motor function and functional skills among young children with cerebral palsy: a systematic review and meta-analysis. BMC Pediatr. 2014 Dec 5;14:292. doi: 10.1186/s12887-014-0292-5. PMID 25475608
- [Background] de Brito Brandao M, Gordon AM, Mancini MC. Functional impact of constraint therapy and bimanual training in children with cerebral palsy: a randomized controlled trial. Am J Occup Ther. 2012 Nov-Dec;66(6):672-81. doi: 10.5014/ajot.2012.004622. PMID 23106987
- [Background] Deppe W, Thuemmler K, Fleischer J, Berger C, Meyer S, Wiedemann B. Modified constraint-induced movement therapy versus intensive bimanual training for children with hemiplegia - a randomized controlled trial. Clin Rehabil. 2013 Oct;27(10):909-20. doi: 10.1177/0269215513483764. Epub 2013 Jul 1. PMID 23818409
- [Background] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924
- [Background] Aarts PB, Jongerius PH, Geerdink YA, van Limbeek J, Geurts AC. Effectiveness of modified constraint-induced movement therapy in children with unilateral spastic cerebral palsy: a randomized controlled trial. Neurorehabil Neural Repair. 2010 Jul-Aug;24(6):509-18. doi: 10.1177/1545968309359767. Epub 2010 Apr 27. PMID 20424191
- [Background] Sakzewski L, Carlon S, Shields N, Ziviani J, Ware RS, Boyd RN. Impact of intensive upper limb rehabilitation on quality of life: a randomized trial in children with unilateral cerebral palsy. Dev Med Child Neurol. 2012 May;54(5):415-23. doi: 10.1111/j.1469-8749.2012.04272.x. Epub 2012 Mar 17. PMID 22429002